CLINICAL TRIAL: NCT02041663
Title: Septic cArdiac Deficiency and MenIngococcal seveRe Sepsis
Acronym: SAMIRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AOR 10106
Record Dates: First submitted 2014-01-20; First posted 2014-01-22 (Estimated); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Meningococcal Infections; Septic Shock; Severe Sepsis
Keywords: brain natriuretic peptide; cardiac function; meningococcal infections; septic shock; severe sepsis
MeSH Terms: conditions — Meningococcal Infections; Shock, Septic; Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Population (Experimental): Repeated brain natriuretic peptide dosages and cardiac echographies up to day 5
  Interventions: Biological: BNP

INTERVENTIONS:
Biological: BNP — Repeated brain natriuretic peptide dosages and cardiac echographies up to day 5

SUMMARY:
Use of brain natriuretic peptide to evaluate the cardiac function in the course of meningococcal septic shock or severe sepsis.

DETAILED DESCRIPTION:
OBJECTIVES: determining sensibility and specificity of BNP blood level to detect myocardial dysfunction in septic shock or severe sepsis due to Neisseria meningitidis in children.

METHODS: Prospective multicentric clinical trial including 7 French pediatric intensive care units. Serial cardiac ultra sounds and blood sampling will be done for patients hospitalized for purpura fulminans beginning at the time of admission in pediatric intensive care. Any child from 6 months to 18 years without preexisting cardiac disease and presenting with purpura fulminans will be enrolled after obtaining consent of both parents. From adult's studies on septic shock and BNP, a total number of 30 patients was calculated to be necessary to prove the interest of BNP in this indication.

ELIGIBILITY:
Inclusion Criteria:

* Children
* 6 months to 18 years aged
* without previous cardiac pathology
* hospitalized in the participating pediatric intensive care units for serious sepsis with extensive purpura

Exclusion Criteria:

* Heart malformative disorder with right-left shunt
* Pre-existent known cardiac insufficiency whatever is the origin
* Concomitant participation in another trial
* Patient in period of exclusion from another trial
* Not membership in a national insurance scheme

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2012-03-05 (Actual); Primary Completion 2018-07-11 (Actual); Study Completion 2018-07-11 (Actual)

PRIMARY OUTCOMES:
Repeated brain natriuretic peptide (BNP) blood level | Up to day 5

SECONDARY OUTCOMES:
Repeated cardiac echography | Up to day 5
PRISM II gravity score | Up to day 5
Organ failure PELOD score | Up to day 5
Troponin rate | Up to day 5
mortality and morbidity (aftereffects) | Day 28 and hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Jean Bergougnoux, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- AP-HP, Necker hospital, Paris, France